CLINICAL TRIAL: NCT01193179
Title: Long-term Co-administration Study of OPC-262 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Phase 3 Study of OPC-262 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262-10-005; JapicCTI-101252 (Other: JAPIC)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-262 (Experimental)
  Interventions: Drug: OPC-262

INTERVENTIONS:
Drug: OPC-262 — Oral administration of tablets for 52 weeks

SUMMARY:
The purpose of this study is to investigate the safety of OPC-262 administered orally in combination with another oral antihyperglycemic agent

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who are capable of giving informed consent
* 2) Patients who are able to take contraceptive measures to avoid pregnancy of the patient or the patient's partner

Exclusion Criteria:

* Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Adverse events, clinical laboratory tests | 52 weeks

SECONDARY OUTCOMES:
Secondary Outcome HbA1c | 52 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Kanto Rigeon
  - Kinki Region
  - Kyushu Region
  - Tohoku Region